CLINICAL TRIAL: NCT05716386
Title: The Effect of Low Salt Diet on CKD Progression:A Randomized Controlled Trial
Brief Title: Effect of Low Salt and Ckd Progression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Collaborators: Science research and innovation (Unknown)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 142/65
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: CKD Progression; Blood Pressure; Proteinuria
Keywords: CKD progression; Low salt; Randomized controlled trial
MeSH Terms: conditions — Proteinuria | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Intervention Model Description: Prospective open labelled randomized controlled trial study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The low sodium diet will be provided low salt diet 1.5 gm/day in three main meals for three months.The food will be provided by the nutritionists and delivered directly to their home
  Interventions: Dietary Supplement: Low salt diet
- Control (Placebo Comparator): The control group will continue with their usual diet and record the food recall
  Interventions: Dietary Supplement: Low salt diet

INTERVENTIONS:
Dietary Supplement: Low salt diet — Low salt diet less than 2 gram per day

SUMMARY:
Whether an intensive short-term dietary sodium restricted intervention will have beneficial effects on the glomerular filtration rate (GFR) and on the susceptibility to develop proteinuria, both measures of kidney function will be the objective of this study

DETAILED DESCRIPTION:
The prevalence of non-communicable disease (NCD including cardiovascular disease (CVD), diabetes mellitus (DM),hypertension(HT) and chronic kidney disease(CKD) continues to rise all over the world and lead to global crisis.The world Health Organization (WHO) shows that more than 50% of the burden of diseases arise from NCD and 30% is attributed to CVD[1] .In Thailand,the prevalence of high blood pressure in population age > 15 is increasing in the past 10 years .In 2022 the HT prevalence was 21.4 and the admission rate of CVD increased from 109.4 to 793.3 per 100,000 population [2]. Cumulating evidence highlights that higher sodium consumption contributes to higher BP [3], thus increasing the risk of cardiovascular disease (CVD) [4,5]. According to the World Health Organization, the restriction of sodium intake to less than 2.3 g/day of sodium corresponding to 5.8 g of salt (or 100 mmol) is one of the most cost-effective measures to improve public health [6]. In particular, in a large cohort study in over 100,000 patients from 18 countries the role of higher salt consumption was associated with increased BP levels [7], and poor CV outcomes [8].In one meta-analysis ,reduce salt intake to 1,800 mg per day will help reduce blood pressure by 2/1 mmHg in non-hypertensive cohorts and 5/2.7 mmHg in hypertensive patients [4].In fact, even minor sodium restriction for only 700-800 mmol/day was associated with reduction of CVD and mortality risks for 20 and 5-7% respectively.

A long-standing line of evidence also shows beneficial effects of salt reduction in patients with chronic kidney disease (CKD) as well as in healthy people [9,10]. A recent review of the evidence for the relationship between salt intake and CKD progression concluded there is consistent evidence to suggest that dietary salt intake is linked with albuminuria and tissue injury [9] [11]. High salt intake is closely associated with the progression of CKD. When the urine sodium-to-creatinine ratio increases by 100 mmol/L, the risk of CKD developing into end-stage renal disease (ESRD) increases by 1.61 times [12,13]. High salt intake leads to renal impairment in various ways, including increasing transforming growth factor (TGF)-β1 production and enhancing oxidative stress and inflammatory response kidney [14-16]. The Lowsalt CKD trial trials had shown that in patients with CKD, salt reduction will have additional beneficial effects on renal effects, reduction of proteinuria,independent of blood pressure lowering effect. reported that salt reduction helped control blood pressure,reduce proteinuria [17] .However,the follow up time was too short. Meta-analysis data from Garofalo et al [18] indicates that low sodium intake ( 4.4 gm/day) in 738 CKD patients from 9 studies significantly reduce systolic blood pressure by 4.9 mmHg (95%CI 6.8/31 mmHg, p <0.001) .The diastolic blood pressure also reduce by 2 mmHg (95%CI 6.8/3.1 mmHg, P<0.001) .In CRIC study[19] which followed a cohort of 3,757 CKD patients for nearly 7 years,the authors found that the high urine sodium group (UNaV > 195 mmoL/day) significantly increased risk for CKD progression and CVD risk. These data support the evidence that reducing dietary sodium can reduce cardiovascular risk and rate of CKD progression.

However, restriction in dietary sodium intake also activates the renin-angiotensin -aldosterone system (RAAS) and sympathetic nervous system[20,21].Low dietary sodium has been reported to be associated with insulin resistance [22]. To date, the connection between sodium intake and CKD progression provided inconsistent results [23]. Although several studies have shown that high dietary sodium intake increases the risk of CKD development or progression [24-26], some results failed to find significant connections to renal outcome [27-30]. In addition, there have also been reports that lower 24-hour urine sodium excretion is associated with higher risk of death and ESRD in individuals with type 1 and type 2 diabetes with overt proteinuria [30,31]. Whether an intensive short-term dietary sodium restricted intervention will have beneficial effects on the glomerular filtration rate (GFR) and on the susceptibility to develop proteinuria, both measures of kidney function will be the objective of this study

ELIGIBILITY:
Inclusion Criteria:

* years with CKD stage 1-3 (estimated glomerular filtration rate (eGFR) of 30-59 ml/min per 1·73 m2
* No recent history of acute illness or hospitalization
* BP >135/85 mmHg or controlled BP with the use of antihypertensive medications.

Exclusion Criteria:

* Serious primary diseases affecting major organs such as the heart, brain, lung, liver, or hematopoietic system
* Active cancers
* Acute infectious diseases
* Pregnancy
* Post solid organs transplantation
* Terminally ill.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Rate of GFR decline | 3 months
  estimeated glomerular filtration rate

SECONDARY OUTCOMES:
Blood pressure status | 3 months
  Blood pressure
Acid-base status | 3 months
  Electrolyte level
Calcium-phosphate balance | 3 months
  calcium,phosphorus level
Proteinuria | 3 months
  24 hour urine protien level

CONTACTS AND LOCATIONS:
Overall Officials: Thananda Trakarnvanich, Principal Investigator — Navamindradhiraj University
Locations (1):
- Faculty of Medicine,Vajira Hospital,Navamindradhiraj University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
We plan to deposit the data to the central repository site such as figshare or Mendeley
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Indefifnitely
Access Criteria: Investigator team member Those who get permission from the principle investigator
URL: https://figshare.com/articles/dataset/datasets/5472970

REFERENCES:
- [Background] Cappuccio FP, Capewell S, Lincoln P, McPherson K. Policy options to reduce population salt intake. BMJ. 2011 Aug 11;343:d4995. doi: 10.1136/bmj.d4995. No abstract available. PMID 21835876
- [Background] Garofalo C, Borrelli S, Provenzano M, De Stefano T, Vita C, Chiodini P, Minutolo R, De Nicola L, Conte G. Dietary Salt Restriction in Chronic Kidney Disease: A Meta-Analysis of Randomized Clinical Trials. Nutrients. 2018 Jun 6;10(6):732. doi: 10.3390/nu10060732. PMID 29882800
- [Background] He J, Mills KT, Appel LJ, Yang W, Chen J, Lee BT, Rosas SE, Porter A, Makos G, Weir MR, Hamm LL, Kusek JW; Chronic Renal Insufficiency Cohort Study Investigators. Urinary Sodium and Potassium Excretion and CKD Progression. J Am Soc Nephrol. 2016 Apr;27(4):1202-12. doi: 10.1681/ASN.2015010022. Epub 2015 Sep 17. PMID 26382905
- [Background] Rhee OJ, Rhee MY, Oh SW, Shin SJ, Gu N, Nah DY, Kim SW, Lee JH. Effect of sodium intake on renin level: Analysis of general population and meta-analysis of randomized controlled trials. Int J Cardiol. 2016 Jul 15;215:120-6. doi: 10.1016/j.ijcard.2016.04.109. Epub 2016 Apr 14. PMID 27111173
- [Background] Graudal NA, Galloe AM, Garred P. Effects of sodium restriction on blood pressure, renin, aldosterone, catecholamines, cholesterols, and triglyceride: a meta-analysis. JAMA. 1998 May 6;279(17):1383-91. doi: 10.1001/jama.279.17.1383. PMID 9582047
- [Background] McQuarrie EP, Traynor JP, Taylor AH, Freel EM, Fox JG, Jardine AG, Mark PB. Association between urinary sodium, creatinine, albumin, and long-term survival in chronic kidney disease. Hypertension. 2014 Jul;64(1):111-7. doi: 10.1161/HYPERTENSIONAHA.113.03093. Epub 2014 Apr 14. PMID 24732890
- [Background] Vegter S, Perna A, Postma MJ, Navis G, Remuzzi G, Ruggenenti P. Sodium intake, ACE inhibition, and progression to ESRD. J Am Soc Nephrol. 2012 Jan;23(1):165-73. doi: 10.1681/ASN.2011040430. Epub 2011 Dec 1. PMID 22135311
- [Background] Mazarova A, Molnar AO, Akbari A, Sood MM, Hiremath S, Burns KD, Ramsay TO, Mallick R, Knoll GA, Ruzicka M. The association of urinary sodium excretion and the need for renal replacement therapy in advanced chronic kidney disease: a cohort study. BMC Nephrol. 2016 Sep 5;17(1):123. doi: 10.1186/s12882-016-0338-z. PMID 27596141
- [Background] Nagata T, Sobajima H, Ohashi N, Hirakawa A, Katsuno T, Yasuda Y, Matsuo S, Tsuboi N, Maruyama S. Association between 24h Urinary Sodium and Potassium Excretion and Estimated Glomerular Filtration Rate (eGFR) Decline or Death in Patients with Diabetes Mellitus and eGFR More than 30 ml/min/1.73m2. PLoS One. 2016 May 2;11(5):e0152306. doi: 10.1371/journal.pone.0152306. eCollection 2016. PMID 27136292
- [Background] Thomas MC, Moran J, Forsblom C, Harjutsalo V, Thorn L, Ahola A, Waden J, Tolonen N, Saraheimo M, Gordin D, Groop PH; FinnDiane Study Group. The association between dietary sodium intake, ESRD, and all-cause mortality in patients with type 1 diabetes. Diabetes Care. 2011 Apr;34(4):861-6. doi: 10.2337/dc10-1722. Epub 2011 Feb 9. PMID 21307382
- [Result] Strong K, Mathers C, Leeder S, Beaglehole R. Preventing chronic diseases: how many lives can we save? Lancet. 2005 Oct 29-Nov 4;366(9496):1578-82. doi: 10.1016/S0140-6736(05)67341-2. PMID 16257345
- [Result] World Health Organization. Country Office for T. Hypertension care in Thailand: best practices and challenges, 2019. Bangkok: World Health Organization. Country Office for Thailand; 2019.
- [Result] He FJ, Li J, Macgregor GA. Effect of longer term modest salt reduction on blood pressure: Cochrane systematic review and meta-analysis of randomised trials. BMJ. 2013 Apr 3;346:f1325. doi: 10.1136/bmj.f1325. PMID 23558162
- [Result] He FJ, MacGregor GA. Salt reduction lowers cardiovascular risk: meta-analysis of outcome trials. Lancet. 2011 Jul 30;378(9789):380-2. doi: 10.1016/S0140-6736(11)61174-4. No abstract available. PMID 21803192
- [Result] Strazzullo P, D'Elia L, Kandala NB, Cappuccio FP. Salt intake, stroke, and cardiovascular disease: meta-analysis of prospective studies. BMJ. 2009 Nov 24;339:b4567. doi: 10.1136/bmj.b4567. PMID 19934192
- [Result] Guideline: Sodium Intake for Adults and Children. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK133309/ PMID 23658998
- [Result] Mente A, O'Donnell MJ, Rangarajan S, McQueen MJ, Poirier P, Wielgosz A, Morrison H, Li W, Wang X, Di C, Mony P, Devanath A, Rosengren A, Oguz A, Zatonska K, Yusufali AH, Lopez-Jaramillo P, Avezum A, Ismail N, Lanas F, Puoane T, Diaz R, Kelishadi R, Iqbal R, Yusuf R, Chifamba J, Khatib R, Teo K, Yusuf S; PURE Investigators. Association of urinary sodium and potassium excretion with blood pressure. N Engl J Med. 2014 Aug 14;371(7):601-11. doi: 10.1056/NEJMoa1311989. PMID 25119606
- [Result] Hooper L, Bartlett C, Davey Smith G, Ebrahim S. Systematic review of long term effects of advice to reduce dietary salt in adults. BMJ. 2002 Sep 21;325(7365):628. doi: 10.1136/bmj.325.7365.628. PMID 12242173
- [Result] Xie X, Atkins E, Lv J, Bennett A, Neal B, Ninomiya T, Woodward M, MacMahon S, Turnbull F, Hillis GS, Chalmers J, Mant J, Salam A, Rahimi K, Perkovic V, Rodgers A. Effects of intensive blood pressure lowering on cardiovascular and renal outcomes: updated systematic review and meta-analysis. Lancet. 2016 Jan 30;387(10017):435-43. doi: 10.1016/S0140-6736(15)00805-3. Epub 2015 Nov 7. PMID 26559744
- [Result] Yuan M, Moody WE, Townend JN. Central blood pressure in chronic kidney disease: latest evidence and clinical relevance. Curr Hypertens Rev. 2014;10(2):99-106. doi: 10.2174/1573402111666141231145931. PMID 25549839
- [Result] Jones-Burton C, Mishra SI, Fink JC, Brown J, Gossa W, Bakris GL, Weir MR. An in-depth review of the evidence linking dietary salt intake and progression of chronic kidney disease. Am J Nephrol. 2006;26(3):268-75. doi: 10.1159/000093833. Epub 2006 Jun 9. PMID 16763384
- [Result] O'Donnell M, Mente A, Rangarajan S, McQueen MJ, Wang X, Liu L, Yan H, Lee SF, Mony P, Devanath A, Rosengren A, Lopez-Jaramillo P, Diaz R, Avezum A, Lanas F, Yusoff K, Iqbal R, Ilow R, Mohammadifard N, Gulec S, Yusufali AH, Kruger L, Yusuf R, Chifamba J, Kabali C, Dagenais G, Lear SA, Teo K, Yusuf S; PURE Investigators. Urinary sodium and potassium excretion, mortality, and cardiovascular events. N Engl J Med. 2014 Aug 14;371(7):612-23. doi: 10.1056/NEJMoa1311889. PMID 25119607
- [Result] Habibi J, Hayden MR, Ferrario CM, Sowers JR, Whaley-Connell AT. Salt Loading Promotes Kidney Injury via Fibrosis in Young Female Ren2 Rats. Cardiorenal Med. 2014 Apr;4(1):43-52. doi: 10.1159/000360866. Epub 2014 Mar 14. PMID 24847333
- [Result] Varagic J, Ahmad S, Brosnihan KB, Habibi J, Tilmon RD, Sowers JR, Ferrario CM. Salt-induced renal injury in spontaneously hypertensive rats: effects of nebivolol. Am J Nephrol. 2010;32(6):557-66. doi: 10.1159/000321471. Epub 2010 Nov 2. PMID 21042014
- [Result] Garg R, Williams GH, Hurwitz S, Brown NJ, Hopkins PN, Adler GK. Low-salt diet increases insulin resistance in healthy subjects. Metabolism. 2011 Jul;60(7):965-8. doi: 10.1016/j.metabol.2010.09.005. Epub 2010 Oct 30. PMID 21036373
- [Result] Anderson CA, Ix JH. Sodium reduction in CKD: suggestively hazardous or intuitively advantageous? J Am Soc Nephrol. 2013 Dec;24(12):1931-3. doi: 10.1681/ASN.2013090923. Epub 2013 Nov 7. No abstract available. PMID 24204000
- [Result] Fan L, Tighiouart H, Levey AS, Beck GJ, Sarnak MJ. Urinary sodium excretion and kidney failure in nondiabetic chronic kidney disease. Kidney Int. 2014 Sep;86(3):582-8. doi: 10.1038/ki.2014.59. Epub 2014 Mar 19. PMID 24646858
- [Result] Dunkler D, Dehghan M, Teo KK, Heinze G, Gao P, Kohl M, Clase CM, Mann JF, Yusuf S, Oberbauer R; ONTARGET Investigators. Diet and kidney disease in high-risk individuals with type 2 diabetes mellitus. JAMA Intern Med. 2013 Oct 14;173(18):1682-92. doi: 10.1001/jamainternmed.2013.9051. PMID 23939297
- [Result] Kieneker LM, Bakker SJ, de Boer RA, Navis GJ, Gansevoort RT, Joosten MM. Low potassium excretion but not high sodium excretion is associated with increased risk of developing chronic kidney disease. Kidney Int. 2016 Oct;90(4):888-96. doi: 10.1016/j.kint.2016.07.012. Epub 2016 Aug 26. PMID 27575557
- [Derived] Trakarnvanich T, Chailimpamontree W, Kantachuvesiri S, Anutrakulchai S, Manomaipiboon B, Ngamvitchukorn T, Suraamornkul S, Trakarnvanich T, Kurathong S. Effect of a Low Salt Diet on the Progression of Chronic Kidney Disease: A Prospective, Open-Label, Randomized Controlled Trial. J Prim Care Community Health. 2024 Jan-Dec;15:21501319241297766. doi: 10.1177/21501319241297766. PMID 39526855